CLINICAL TRIAL: NCT05915299
Title: US National OCS Heart Perfusion (OHP) Registry
Status: Recruiting | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-HEART-OHP-II
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Heart Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- OCS Heart Transplant Recipients: All heart transplant recipients who are transplanted with an OCS perfused donor heart are eligible for this registry.
  Interventions: Device: OCS Heart

INTERVENTIONS:
Device: OCS Heart — The TransMedics® Organ Care System (OCS) Heart System is an FDA approved portable extracorporeal heart perfusion and monitoring system.
  The OCS Heart System's innovative technology was designed to comprehensively overcome the historical limitations of cold storage. The OCS Heart System expands the utilization of donor hearts by enabling the use of donor hearts deemed unsuitable for procurement and transplantation at initial evaluation due to limitations of cold static cardioplegic preservation.

SUMMARY:
This Registry is a sponsor initiated, multi-center, observational post-approval registry with independent academic oversight.

DETAILED DESCRIPTION:
The objective of this US National OHP Registry is to collect data on the post-transplant clinical outcomes of all donor hearts preserved and assessed on the OCS Heart System and to document the performance of the OCS Heart device in the real-world setting after FDA approval in the US.

The US National OHP Registry will enroll all heart transplant recipients who are transplanted with an OCS-perfused donor heart in the Registry. Patients' clinical outcomes will be followed up to five years post-transplant, loss to follow up, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All heart transplant recipients who are transplanted with an OCS perfused donor heart are eligible for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2033-08-31 (Estimated)

PRIMARY OUTCOMES:
Recipients' patient and graft survival | Up to 5 years post-transplant
  Recipients' patient and graft survival rates will be the primary clinical outcomes measures for all OCS Heart transplanted recipients compared to recipients receiving heart transplants using non-OCS preservation methods (cold static storage or other perfusion devices or a combination of both). This data will be obtained directly from UNOS/OPTN database.

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Stanford University, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Boulder, Boulder, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford, Detroit, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mount Sinai, New York, New York
  - Columbia University Irving Medical Center/ New York Presbyterian Hospital, New York, New York
  - Montefiore, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Scott and White, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University Health, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Aurora St Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin